CLINICAL TRIAL: NCT01011283
Title: A Randomized, Open-label, Parallel-Group Study Comparing the Efficacy and Safety of DACOGEN (Decitabine) for Injection and VIDAZA (Azacitidine) for Injection In Subjects With Intermediate or High Risk Myelodysplastic Syndromes (MDS)
Brief Title: To Demonstrate Superiority of Decitabine Over Azacitidine in Subjects With Intermediate- or High-risk MDS.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped due to insufficient enrollment.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7373-A001-401
Record Dates: First submitted 2009-11-05; First posted 2009-11-11 (Estimated); Results first posted 2013-09-18 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS; Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine; Azacitidine

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: decitabine
- 2 (Active Comparator)
  Interventions: Drug: azacitidine

INTERVENTIONS:
Drug: decitabine — decitabine 20 mg/m^2 /day intravenous (IV) infusion for 5 days every 28 days
  Other Names: Dacogen (decitabine)
  Arms: 1
Drug: azacitidine — azacitidine 75 mg/m^2 /day subcutaneous (SC) injection for 7 days every 28 days
  Other Names: Vidaza (azacitidine)
  Arms: 2

SUMMARY:
The purpose of this study is to compare the response of patients with Intermediate or High Risk myelodysplastic syndromes (MDS) following treatment with decitabine or azacitidine.

ELIGIBILITY:
Inclusion Criteria

Subjects who meet all of the following criteria may be included in the study:

1. Must have a diagnosis of primary myelodysplastic syndromes (MDS) of Intermediate-1 transfusion dependent, Intermediate-2, or High-risk [defined by International Prognostic Scoring System (IPSS) score of ≥0.5] and recognized French-American-British (FAB) classifications
2. Male or female, 18 years of age or older with signed informed consent
3. Adequate renal function
4. Demonstrated normal liver function
5. Female subjects of childbearing age must have negative pregnancy test within 1 week of study entry and agree to use adequate contraception for the duration of the trial and for a minimum of six months after last dose of decitabine or azacitidine received.
6. Male subjects must agree to use adequate contraception for the duration of the trial and for a minimum of six months after last dose of decitabine or azacitidine received.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Current use of radiotherapy for extramedullary disease for 2 weeks prior to entering study (permitted if > 2 weeks from study entry and if recovered from toxic effects of therapy)
2. Systemic fungal, bacterial, or viral infection which is not controlled (i.e., ongoing signs or symptoms of infection and without improvement despite appropriate treatment)
3. Pregnancy or current lactation
4. Significant concurrent disease, illness, or psychiatric disorder
5. Treatment with an investigational agent 30 days prior to the first dose of decitabine or azacitidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Stein, Study Director — Eisai Inc.
Locations (19):
- United States (19):
  - Birmingham Hematology and Oncology Associates, Birmingham, Alabama
  - Stanford University Cancer Center, Stanford, California
  - Stockton Hematology Oncology, Stockton, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Pasco Pinellas Cancer Center, New Port Richey, Florida
  - Gulf Coast Oncology, St. Petersburg, Florida
  - University of Chicago, Chicago, Illinois
  - Siouxland Haeatology - Oncology Associates, Sioux City, Iowa
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Sletten Cancer Institute, Great Falls, Montana
  - Cornell Medical Center, New York, New York
  - Carolinas Medical Center NorthEast NorthEast Oncology Associates, Concord, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Oncology and Hematology Care, Cincinnati, Ohio
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Gunderson Clinic Ltd., La Crosse, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 20 centers in U.S. during the period of Feb 2010 to Jan 2011.
Groups:
- Decitabine 20 mg/m^2: decitabine : decitabine 20 mg/m^2 /day intravenous (IV) infusion for 5 days every 28 days
- Azacitidine 75 mg/m^2: azacitidine : azacitidine 75 mg/m^2 /day subcutaneous (SC) injection for 7 days every 28 days
Period: Overall Study
Arm/Group | Decitabine 20 mg/m^2 | Azacitidine 75 mg/m^2
Started | 13 | 13
Completed | 2 | 2
Not Completed | 11 | 11
Not completed — Adverse Event | 4 | 2
Not completed — Progressive Disease | 0 | 2
Not completed — Terminated by Sponsor | 5 | 5
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decitabine 20 mg/m^2 | Azacitidine 75 mg/m^2 | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (11.60) | 70.8 (9.13) | 72.3 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 12 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR), Defined as Proportion of Patients Having Complete Response (CR) and Marrow Complete Response (mCR) After Completion of 3 Cycles of Study Drug.
Description: Based on Modified International Working Group Response Criteria for Altering Natural History of Myelodysplastic Syndromes.
  Complete Response: Bone marrow: ≤ 5% myeloblasts with normal maturation of all cell lines. Persistent dysplasia will be noted. Peripheral blood Hgb ≥ 11 g/dL; Platelets ≥ 100 X 10^9/L; Neutrophils ≥ 1.0 X 10^9/Lb; Blasts 0%.
  Marrow Complete Response: Bone marrow: ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment. Peripheral blood: if hematological improvement responses, they will be noted in addition to marrow CR.
Time Frame: 13 Weeks
Population: Intent to Treat Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Decitabine 20 mg/m^2 | Azacitidine 75 mg/m^2
Number analyzed (Participants) | 11 | 12
Percentage of Participants
  Overall Response Rate | 0 | 0
  Complete Response | 0 | 0
  Marrow Complete Response | 0 | 0
  Partial Response | 0 | 0
  Stable Disease | 45.5 | 25.0

2. Secondary Outcome: Overall Response Rate (ORR), Defined as Proportion of Patients Having Complete Response (CR) and Marrow Complete Response (mCR) After Completion of 6 Cycles of Study Drug.
Description: as for outcome 1
Time Frame: 36 Weeks
Population: Intent to Treat Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Decitabine 20 mg/m^2 | Azacitidine 75 mg/m^2
Number analyzed (Participants) | 11 | 12
Percentage of Participants
  Overall Response Rate | 9.1 | 8.3
  Complete Response | 9.1 | 8.3
  Marrow Complete Response | 0 | 0
  Partial Response | 9.1 | 0
  Stable Disease | 36.4 | 16.7

ADVERSE EVENTS:
Arm/Group | Decitabine 20 mg/m^2 | Azacitidine 75 mg/m^2
Serious Adverse Events (participants affected / at risk) | 7/13 | 7/13
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine 20 mg/m^2 (N=13) | Azacitidine 75 mg/m^2 (N=13)
Pancytopenia (Blood and lymphatic system disorders) | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Cardiac disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0
Aspergillosis (Infections and infestations) | 1 | 0
Neutropenia sepsis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine 20 mg/m^2 (N=13) | Azacitidine 75 mg/m^2 (N=13)
Anemia (Blood and lymphatic system disorders) | 7 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 4 | 3
Neutropenia (Blood and lymphatic system disorders) | 6 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 5
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 2 | 0
Erythema of eyelid (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 0 | 2
Eye pain (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 3
Diarrhea (Gastrointestinal disorders) | 4 | 5
Fecal incontinence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 9
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 8
Asthenia (General disorders) | 1 | 2
Catheter site erythema (General disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 0
Chills (General disorders) | 2 | 1
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 5 | 7
Feeling jittery (General disorders) | 0 | 1
Injection site erythema (General disorders) | 0 | 4
Injection site hemorrhage (General disorders) | 0 | 1
Injection site edema (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 3
Injection site rash (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 4
Nodule (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Edema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Acute sinusitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 2 | 0
Paronchia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 2
Contusion (Infections and infestations) | 1 | 1
Post procedural discharge (Infections and infestations) | 0 | 1
Skin laceration (Infections and infestations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Breath sounds abnormal (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 3
Memory impairment (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2
Mental status changes (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No